CLINICAL TRIAL: NCT04067973
Title: Impact of Prematurity on the Morphological and Tomographic Aspect of the Papilla
Brief Title: Impact of Prematurity on the Optic Nerve
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0026
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Ocular Surface Disease; Premature
Keywords: optic nerve; premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: Premature subjects benefit from the examinations described in the protocol, namely automated refractometry, intraocular air pressure, biometrics (with axial length and pachymetry (corneal thickness) performed by the same machine at the same time), a photo of the fundus (retinophotography) and an OCT RNFL. These examinations are necessary for the follow-up of premature children.
  All children examined at Nantes University Hospital benefit systematically from: automated refractometry, intraocular pressure in the air and a photo of the fundus.
- control: controls benefit from two additional tests: RNFL OCT and biometrics. The duration of the RNFL OCT is about 2 minutes, with a total of 10 seconds per eye, the rest being computer manipulation.
  The biometrics take about 2 minutes to complete, with a total of 30 seconds per eye, the rest being computer manipulation.
  These two reviews are conducted on the same day as the initial consultation and directly following the consultation.

SUMMARY:
The purpose of this protocol is to study the consequences of prematurity on the optic nerve. Indeed, the work already carried out on the subject suggests that prematurity induces suffering of the optic nerve with a loss of optical fibre, an essential element in the transmission of the visual nerve signal to the brain.

The investigators will therefore study two populations: a population of premature infants aged 5 to 10 years, and a control population of term infants.

The examinations performed are painless, non-invasive and non-irradiating. To date, there are no known adverse reactions to these tests. These examinations are a photo of the fundus (retinophotography), a pachymetry (measurement of the thickness of the non-contact cornea), an OCT RNFL (optical coherence tomography, scanner of the non-irradiating non-painful optical nerve) and the taking of the IOP (intraocular pressure).

They aim to measure the main morphological characteristics of the eye and the optic nerve.

This is a prospective observational study. The inclusion and measurements necessary for the study are made on the day of the consultation.

The expected results will provide new data on this population of premature infants, allowing for better management if a pathology involving the optic nerve were to occur at any age in these patients.

DETAILED DESCRIPTION:
The prematurity of the newborn is now a major theme in medical research. Indeed, technological progress makes it possible to revive increasingly premature children. But being born premature also brings many complications, some of which are already well known (pulmonary, cardiac, digestive complications, etc....). At the ophthalmological level, the retinopathy of the premature child is an entity already well described, this retinal vascularization anomaly leads to many complications on the child's visual future. The optic nerves of premature infants are described as larger than those of normal children.

Recently, a new ophthalmological condition has been described. This is the damage to the optic nerve of the premature baby, characterized by a loss of optical fibres, of major importance in the transmission of the visual signal to the brain.

The aim of this study is to characterize the particularities of the optic nerve of the premature child, as there is currently very little data available on it in this context. Some studies have reported this, but with results that are not always homogeneous. For example, some studies report a lack of optic fiber in the temporal area of the optic nerve, while others find more pronounced atrophy on the nasal side, which has practical consequences in the examination and monitoring of these children.

A better understanding of these disorders would make it possible to establish monitoring protocols for these children born with nerve fibre deficiency, especially to prevent subsequent fibre loss due to any pathology of ocular tone, the best known of which is glaucoma.

The purpose of this prospective study is to compare the aspects of optic nerves in premature infants compared to those of optic nerves in non-premature infants. This aspect changes with age, with a progressive physiological decrease in the thickness of optic fiber within the optic nerve over time. It is therefore essential to match the two age groups to exploit this data.

ELIGIBILITY:
Inclusion Criteria:

* For patients:
* between 5 and 10 years old
* Premature births: before 37 weeks of amenorrhea
* To be able to benefit from the examinations necessary for the study (being able to set a target, to install correctly on the machines)

For control:

* Aged between 5 and 10 years old
* Born after 37 SA
* No known ophthalmological pathologies
* To be able to benefit from the examinations necessary for the study (being able to set a target, to install correctly on the machines)

Exclusion Criteria:

* Patients who cannot benefit from the examinations (patients in wheelchairs, whose psychomotor delay prevents a good understanding of the examination and the need to set a target)
* patient under the protection of justice.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Prospective monocentric case-control study, based on the use of data recovered after a single patient visit.
  Conduct of a visit for the patient (case control):
  * Reception of the patient and his parents or legal representatives
  * Information to the patient and his parents or legal representatives of the study
  * Carrying out the standard consultation (optical correction most often) then carrying out additional examinations necessary for the study.
  * This visit is unique, there will be no further visits.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-02 (Estimated); Primary Completion 2020-03-02 (Estimated); Study Completion 2020-09-02 (Estimated)

PRIMARY OUTCOMES:
Compare the thickness of the optical fibres measured in OCT RNFL between premature subjects and controls. | 10 minutes
  The examinations performed are painless, non-invasive and non-irradiating. To date, there are no known adverse reactions to these tests. These examinations are a photo of the fundus (retinophotography), a pachymetry (measurement of the thickness of the non-contact cornea), an OCT RNFL (optical coherence tomography, scanner of the non-irradiating non-painful optical nerve) and the taking of the IOP (intraocular pressure).
  They aim to measure the main morphological characteristics of the eye and the optic nerve.
  We will therefore study two populations: a population of premature infants aged 5 to 10 years, and a control population of term infants.

SECONDARY OUTCOMES:
Compare the cup/disc ratio | 20 seconds
  Compare the cup/disc ratio (optic nerve excavation, a criterion well used in the study of glaucoma) between the premature population and the control population.
eye length | 10 seconds
  compare the measurement of the axial eye length (eye length) between the two populations.
Intraocular tension | 20 seconds
  compare the intraocular tension (which can lead to a loss of optical fibre if too high, a criterion measured to avoid any bias induced by hypertonia on the thickness of the optical fibres) between the two populations.
Pachymetry | 20 seconds
  compare pachymetry (corneal thickness, measurement that may interfere with intraocular pressure measurement) between premature born patients and controls
refractive measurements | 20 seconds
  compare refractive measurements (myopia, hyperopia, astigmatism) between the two populations